CLINICAL TRIAL: NCT00002778
Title: GRANULOCYTE-MACROPHAGE COLONY STIMULATING FACTOR (Rhu-GM-CSF) FOR REDUCTION OF LEUKEMIC RELAPSE AFTER T-LYMPHOCYTE DEPLETED ALLOGENEIC BMT FOR CHRONIC MYELOID LEUKEMIA
Brief Title: Sargramostim Following Allogeneic Bone Marrow Transplantation in Treating Patients With Chronic Myelogenous Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: subject accrual and data analysis is completed.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000064783; P01CA015396 (NIH); P30CA006973 (NIH); JHOC-J9449; BRLX-001.0649; JHOC-94110404; NCI-V96-0900
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-04

CONDITIONS: Leukemia
Keywords: relapsing chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; Philadelphia chromosome positive chronic myelogenous leukemia; Philadelphia chromosome negative chronic myelogenous leukemia; atypical chronic myeloid leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative | interventions — sargramostim

INTERVENTIONS:
Biological: sargramostim
Biological: therapeutic allogeneic lymphocytes
Procedure: allogeneic bone marrow transplantation
Procedure: in vitro-treated bone marrow transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with allogeneic bone marrow transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells. Colony-stimulating factors such as sargramostim may increase the number of immune cells found in bone marrow or peripheral blood, and may help a person's immune system recover from the side effects of chemotherapy.

PURPOSE: Phase II trial to study the effectiveness of allogeneic bone marrow transplantation followed by sargramostim in treating patients who have chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether the use of sargramostim (GM-CSF) after T-cell depleted, CD34-positive cell-supplemented allogeneic bone marrow transplantation can reduce leukemic relapse in patients with chronic myelogenous leukemia.

OUTLINE: Patients receive myeloablation with busulfan and cyclophosphamide on an approved protocol. Allogeneic bone marrow is harvested and treated in vitro with anti-CD34 antibody. T-cell depleted, CD34-positive cell-supplemented bone marrow is infused on day 0. Patients receive high-dose sargramostim (GM-CSF) subcutaneously (SC) beginning on day 5 and continuing until blood counts recover and then low-dose GM-CSF SC continuing until day 60.

Donor lymphocyte infusions or second unmodified allogeneic bone marrow transplantation without GM-CSF is considered in case of primary or secondary engraftment failure.

Patients are followed every month for 3 months, every 3 months for 1 year, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study within approximately 6-10 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of chronic myelogenous leukemia (CML) documented by cytogenetic and molecular analyses at Johns Hopkins

  * Philadelphia chromosome (Ph)-positive or -negative CML

    * Ph-negative CML allowed with presence of either:

      * BCR-ABL rearrangement (on molecular, fluorescent in situ hybridization, or polymerase chain reaction analyses)
      * p210 protein
* One of the following:

  * Patient age 18 to 65
  * Disease duration longer than 3 years
  * Accelerated phase CML
* Accelerated phase diagnosis based on any of the following:

  * More than 10% to less than 30% blasts in blood or bone marrow
  * No hematologic response to prior conventional therapy (hydroxyurea or interferon)
  * Extramedullary disease (e.g., progressive splenomegaly or lymphadenopathy)
  * Basophilia greater than 10% in blood or bone marrow
  * Other cytogenetic abnormalities in addition to a single Ph chromosome
  * Second chronic phase
* Failure on interferon suggested of patients over age 18 with chronic phase CML, with failure defined as:

  * No detectable Ph-negative metaphases in marrow after 6 months
  * No progressive increase in Ph-negative metaphases in marrow after 6-12 months
  * Less than 50% Ph-negative metaphases after 1 year
  * No complete cytogenetic remission after 2 years
  * Intolerance to interferon therapy
* No blast crisis CML, chronic myelomonocytic leukemia, or juvenile CML
* The following conditions are allowed:

  * Leukocyte count abnormalities
  * Fibrosis
  * Anemia
  * Fever or bone pain
  * Thrombocytopenia
  * Bone marrow reticulin
* Availability of an HLA-identical sibling donor

  * At least 3 years of age (priority given to donors over age 10)
  * Priority given to CMV-negative donor if patient CMV-negative
  * No medical or psychiatric condition that precludes transplant procedure

PATIENT CHARACTERISTICS:

Age

* 18 to 65

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics

Hepatic

* Not specified

Renal

* Not specified

Other

* No history of intolerance to sargramostim (GM-CSF)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 1995-02; Primary Completion 2005-02 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: B. Douglas Smith, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States